CLINICAL TRIAL: NCT05586828
Title: A Single-center Retrospective Cohort Study to Explore the Prognostic Significance of CONUT in Elderly With HFpEF and Compare Controlling Nutritional Status Score With Other Objective Nutritional Indices. The Primary Endpoint of This Study Was Readmission Due to HF and All-cause Mortality in 1 Year After Hospitalization.
Brief Title: A Single-center Retrospective Cohort Study to Explore the Prognostic Significance of CONUT in Elderly CAD Patients With HFpEFand Compare CONUT With Other Objective Nutritional Indices.
Status: Completed | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BeijingTH20210812chz1
Record Dates: First submitted 2022-10-17; First posted 2022-10-19 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2022-05

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Malnutrition; Aged; Prognosis
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- different controlling nutritional status score

SUMMARY:
HF is an advanced or terminal stage of various heart diseases, with high rehospitalization and mortality rates. In HF patients, undernutrition is not uncommon and represents one of the most significant determinants of poor clinical outcomes. Therefore, nutritional management is of paramount importance for patients with HF.The basic method of nutritional management is to effectively identify the nutritional status of patients with heart failure, especially in elderly patients with heart failure who are not easy to find in the early stage. Limited data are available regarding the association between CONUT score and prognosis in elder patients with HFpEF, despite its easy availability in routine blood chemistry. Therefore, we aimed to evaluate the prognostic significance of CONUT score and to compare it with other well-established nutritional indices in HFpEF, a common HF phenotype in the elderly population with coronary artery disease.

This was a single-center retrospective cohort study which were approved by the Clinical Research Ethics Committee of our hospital (TRECKY2021-185). Written informed consent was obtained from all patients.

Participants were accorded with diagnostic criteria of CAD and HFpEF excluding rheumatic heart disease, congenital heart disease, acute myocardial infarction, hemodialysis or hemofiltration, tumour activity, urgent surgery, death during hospitalization, HF of unknown reasons, New York Heart Association(NYHA) class1and data deficiency. Demographic characteristics and medical parameters were collected from the electronic medical record system . All enrolled patients were followed-up in an outpatients setting. The primary endpoint of this study was readmission due to heart failure and all-cause mortality in the first year after hospitalization. To explore the prognostic significance of controlling nutritional status score in elderly with ejection fraction preserved heart failure and compare controlling nutritional status score with other objective nutritional indices.All analyses were performed using Statistical Product Service Solutions(SPSS) version 19.0 .

ELIGIBILITY:
Inclusion Criteria:

1. Elderly patients (≧65years old) were accorded with diagnostic criteria of coronary artery disease, HFpEF and NYHA Ⅱ-Ⅳ
2. Coronary artery disease was defined
3. The diagnosis of HF was made according to the recommendations of the European Society of Cardiology .
4. HFpEF was defined
5. Severity of functional class was based on NYHA scale.

Exclusion Criteria:

1. Rheumatic heart disease
2. congenital heart disease
3. acute myocardial infarction
4. hemodialysis or hemofiltration
5. tumour activity, urgent surgery
6. death during hospitalization
7. HF of unknown reasons
8. NYHA classⅠ
9. data deficiency
10. loss of follow-up

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly HFpEF Ⅱ-Ⅳ patients with coronary heart disease hospitalized in the Department of Geriatrics Medical Department of Beijing Tongren Hospital affiliated to Capital Medical University from January 1, 2017 to December 31, 2019 were selected
Sampling Method: Non-Probability Sample
Enrollment: 780 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
readmission due to heart failure in the first year after hospitalization | up to one year
all-cause mortality in the first year after hospitalization | up to one year

CONTACTS AND LOCATIONS:
Overall Officials: YING CHEN, Chief Physician, Study Chair — Beijing Tongren Hospital; HUI ZHENG, M.D., Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Chen Y, Zheng H, He Y. Prognostic significance of controlling nutritional status in older adults with heart failure with preserved ejection fraction: a prospective comparative study with other objective nutritional indices. Aging Clin Exp Res. 2023 Jun;35(6):1305-1315. doi: 10.1007/s40520-023-02395-x. Epub 2023 Apr 1. PMID 37005959